CLINICAL TRIAL: NCT05217017
Title: Psychometric Validation of the French Version of the Fear Avoidance Component Scale (FACS)
Brief Title: French Version of Fear-Avoidance Component Scale (FACS-FR)
Acronym: FACS-Fr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Guillaume Léonard, Professor, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-4356b
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Kinesiophobia; Chronic Pain
Keywords: Kinesiophobia; Chronic Pain; Fear-avoidance
MeSH Terms: conditions — Kinesiophobia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic pain (Experimental): Fear-avoidance components scale
  Interventions: Diagnostic Test: FACS

INTERVENTIONS:
Diagnostic Test: FACS — Diagnostic Test: Assessment of disability and behavior (by questionnaires)

SUMMARY:
Chronic musculoskeletal disorders are global burden for economy. Fear-avoidance (FA) seems be a predictor for the transition from subacute to chronic pain. One of the most famous scales to access FA is the Tampa scale of kinesiophobia, but several responders think some items are not clear, too narrow or too general. A new scale, the Fear-Avoidance Components Scale (FACS) was developed by Neblett et al. in 2015 to assess FA. It is a comprehensive set of concepts that more effectively addresses all the essential issues of the FA concept than the current scales. The new scale comprehensively assesses all cognitive, emotional, and behavioral components related to the updated FA model by combining items from well-known scales in the context of the FA model with items on perceived injury-related victimization and blame. A French version of the FACS is currently lacking. The aim of this study is to provide a translation and validation of a French version of FACS in patients with musculoskeletal disorders.

DETAILED DESCRIPTION:
The process is done in two steps to allow the achievement of our two study objectives (translation and validation), with two different cohorts of patients.

First, for the French translation of the FACS, a pre-test with a first cohort of 30 patients will be performed. These patients will have to fill in the French version of the paper questionnaire and answer a second one on their interpretation and understanding of the questions. Each question will be evaluated by the patient. A report will be made with the patients' answers to the questionnaire and reported to the translation committee, then modifications will be made to the translation if necessary. If changes are made, a second pre-test will be done until no changes are needed.

In a second phase, once the French version is finalized, the second cohort of 50 patients will follow the patient schedule presented in Table I. In more detail, at the initial consultation, the diagnosis of chronic pain should be made by the center's orthopedist. At the same time, the orthopedist, resident, or research assistant will validate, through free and informed consent, whether or not the patient agrees to participate in the study, i.e., T0. At this T0, the patient will have to fill out the four questionnaires, which are FACS, Tampa scale for kinesiophobia French Canadian version (EKT-CF), Pain catastrophizing scale French Canadian version (PCS-CF) and Hospital anxiety and depression scale French version (HADS). The questionnaires will be completed in paper form.

At T1, i.e. seven days later, the patient will have to take the FACS French version again on the REDcap platform. This time frame is short enough to allow for a similar or even identical state of function as at T0 for the assessment of test-retest reliability. Patients with a significant change in status will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Current chronic pain complaint is not surgically treated (at least 6 weeks of pain)
* Not being currently treated by a physiotherapist for pain complaint
* French language is mother tongue

Exclusion Criteria:

* Pain from a non-musculoskeletal origin (e.g., tumour)
* Neurological disease
* Impaired cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
FACS | day 0
  The fear-avoidance component scale evaluating fear-avoidance (for all participants) 20 items range from 0-100
FACS | day 7
  The fear-avoidance component scale evaluating fear-avoidance (for all participants) 20 items range from 0-100
TSK | day 0
  Questionnaire evaluating kinesiophobia (for all participants) 17 items total score from 17-68
PCS | day 0
  Pain catastrophizing scale (for all participants) 13 items total score from 0-52
HADS | day 0
  Hospital anxiety and depression scale is a questionnaire evaluating anxiety and depression (for all participants) 2 subscales: anxiety (7 items) and depression (7 items) Total score 0-21 per subscale

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Leonard, Pr, Study Director — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS (CRCHUS), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No